CLINICAL TRIAL: NCT01385176
Title: Neural Cardiac Therapy for Heart Failure Study
Brief Title: Neural Cardiac Therapy for Heart Failure Study (NECTAR-HF)
Acronym: NECTAR-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NECTAR-1109
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Congestive Heart Failure
Keywords: Heart failure; Congestive heart failure; New York Heart Association Class II-III; Vagal therapy; Vagal nerve stimulation
MeSH Terms: conditions — Heart Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Patients were randomized in a 2:1 ratio to receive therapy (VNS ON) or control (VNS OFF) for a 6-month period. The primary endpoint was the change in LVend systolic diameter (LVESD) at 6 months for control vs. therapy, with secondary endpoints of other echocardiography measurements, exercise capacity, quality-of-life assessments, 24-h Holter, and circulating biomarkers.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapy (Experimental): Implant of investigational device system for vagus nerve stimulation. Patients were randomized in a 2 : 1 ratio to receive therapy (VNS ON) or control (VNS OFF) for a 6-month period.
  The experimental arm was receiving vagus nerve stimulation during the first 6 months after implant.
  Titration during the randomization phase with delivery of highest tolerable by patient stimulation current.
  Blood Draw before implant and 6 months after implant. Titration after the randomization phase with adjustments of the chronically highest tolearble by patient current.
  Interventions: Device: Implant of investigational device system; Procedure: Titration during the randomization phase; Procedure: Titration after the randomization phase; Diagnostic Test: Blood Draw
- Control (Sham Comparator): Implant of investigational device system for vagus nerve stimulation. Control group was implanted with study system like the experimental arm, but was not receiving experimental vagus nerve stimulation therapy during the first 6 months after implant. 6-month after implant a cross-over took place and the control arm also started to receive experimental vagus nerve stimulation.
  Blood Draw before implant and 6 months after implant. Titration after the randomization phase with adjustments of the chronically highest tolearble by patient current.
  Interventions: Device: Implant of investigational device system; Procedure: Titration after the randomization phase; Diagnostic Test: Blood Draw

INTERVENTIONS:
Device: Implant of investigational device system — Vagus nerve stimulation lead was wrapped around the right cervical vagus nerve and then connected to a stimulator permanently implanted in the right pectoral region.
Procedure: Titration during the randomization phase — Amplitude of the chronically delivered vagus nerve stimulation in the experimental arm was adjusted to the highest tolerable by patient value. No chronically delivered vagus nerve stimulation in the control arm during the randomization phase.
  Arms: Therapy
Procedure: Titration after the randomization phase — Amplitude of the chronically delivered vagus nerve stimulation was adjusted to the highest tolerable by patient value in all patients in both arms of the study.
Diagnostic Test: Blood Draw — Blood draw before implant and 6 months after implant at the end of the randomization phase.

SUMMARY:
The NECTAR-HF feasibility trial is designed to evaluate the application of right vagal nerve stimulation in heart failure patients with a New York Heart Association Class III, an ejection fraction equal to or less than 35 %, and a narrow QRS duration equal to or less than 130 ms.

DETAILED DESCRIPTION:
The objectives of this study are to assess the impact of right vagal nerve stimulation on left ventricular remodeling, functional capacity, quality of life, and other measures in heart failure patients over a 6-month period. In addition, the study will assess the safety of the NECTAR-HF study system over an 18-month period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above, and of legal age to give informed consent specific to national laws
* Willing and capable of providing informed consent
* Capable of participating in all testing associated with this clinical investigation
* Stable symptomatic heart failure NYHA class II-III
* Left ventricular (LV) ejection fraction equal or smaller than 35 %
* Left ventricular end diastolic diameter (LVEDD) of 5.5 cm or greater
* Prescribed to optimal pharmacologic therapy

Exclusion Criteria:

* QRS larger than 130 ms
* Patients who have been hospitalized for heart failure and who required the use of HF IV therapy within 30 days before enrollment
* Patients unable to tolerate anesthesia required for implant
* Patients with unstable angina, myocardial infarction, PTCA, coronary artery bypass graft, cerebral vascular accident, or transient ischemic attack within previous 90 days before enrollment
* Patients whose primary cause of heart failure is mitral or aortic valve disease, with a severe classification
* Patients with persistent or permanent atrial fibrillation within 90 days prior to enrollment
* Pacemaker indicated patients
* Patients whose heart failure is due to congenital heart disease
* Patients who have started treatment for sleep apnea or sleep disordered breathing with therapies to maintain airway patency (e.g., CPAP, Bi-PAP,APAP) with or without oxygen supplementation within the previous 6 months prior to enrollment
* Patients with hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g. amyloidosis, sarcoidosis)
* Patients with documented chronic obstructive lung disease
* Patients on or indicated for renal dialysis
* Type 1 diabetic patients
* Type 2 diabetic patients that have been treated with insulin for more than 5 years prior to enrollment
* Patients with a life expectancy of less than 12 months per physician judgment
* Patients involved in any concurrent clinical investigation
* Women of childbearing potential who are or might be pregnant at the time of the study or breastfeeding
* Patients with a prior cardiac transplant or expecting a heart transplant operation within the next 12 months
* Patients with a prior vagotomy
* Patients with prior or existing vagal nerve stimulation treatment
* Patients implanted with any active implantable medical device other than a left sided single or dual chamber implantable cardioverter defibrillator (ICD) with bipolar sensing, or a left sided CRT device with each sensing channel programmed to either bipolar sensing or no sensing. All CRT patients must have had CRT for at least 1 year prior to enrollment. The total number of CRT patients will not exceed 30
* Patients with locally implanted semi-/permanent devices such as vascular catheters, etc. that would interfere with the NECTAR-HF study system
* Patients with previously implanted devices on the right side that became infected before removal
* Patients with previous neck surgery and resultant scar formation that interferes with the ability to implant the study system on the right side of the neck (Thyroid/parathyroid, carotid artery etc)
* Patients with known recurrent nerve paralysis
* Patients who have undergone radiotherapy for thyroid disease/cancer
* Patients who have existing or prior tracheotomy
* Patients with severe vertebral cervical disease and limited mobility in the neck; includes those that frequently wear a brace
* Patients with carotid murmur/vascular bruit/carotid artery lesion
* Patients with known/suspected vascular malformation in carotid/vertebral circulatory bed
* Patients who are likely to need an MRI of the neck area because of previous medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-09-21 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Faiez Zannad, M.D., Principal Investigator — Centre d'Investigation Clinique (CIC), Batiment Louis Mathieu, CHU de Nancy
Locations (21):
- UCL Bruxelles, Brussels, Belgium
- Nemocnice Na Homolce, Prague, Czechia
- France (2):
  - Centre d'Investigation Clinique Pierre Drouin, CHU de Nancy, Vandœuvre-lès-Nancy, Nancy
  - CHRU de Lille - Hôpital Cardiologique, Lille
- Germany (4):
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau bei Berlin, Brandenburg
  - Universitätsmedizin Göttingen, Göttingen
  - Universitäres Herzzentrum GmbH, Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Leipzig, Leipzig
- Italy (3):
  - Azienda Ospedaliera Niguarda Cà Granda, Milan
  - A. O. Dei Colli - Monaldi, Napoli
  - Policlinico San Matteo, Pavia
- Netherlands (2):
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - UMC Utrecht, Utrecht
- Spain (3):
  - Clínica Universitaria de Navarra, Avenida Pio XII s/n, Pamplona, Navarre
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Doce de Octubre, Madrid
- United Kingdom (5):
  - University Hospitals Bristol, NHS Foundation Trust, Bristol, England
  - Liverpool Heart and Chest Hospital, NHS Foundation Trust, Liverpool, England
  - The Heart Hospital, University College London Hospitals, NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust, St. Mary's Hospital, London, England
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Ferrari GM, Tuinenburg AE, Ruble S, Brugada J, Klein H, Butter C, Wright DJ, Schubert B, Solomon S, Meyer S, Stein K, Ramuzat A, Zannad F. Rationale and study design of the NEuroCardiac TherApy foR Heart Failure Study: NECTAR-HF. Eur J Heart Fail. 2014 Jun;16(6):692-9. doi: 10.1002/ejhf.80. Epub 2014 May 20. PMID 24846173
- [Result] Zannad F, De Ferrari GM, Tuinenburg AE, Wright D, Brugada J, Butter C, Klein H, Stolen C, Meyer S, Stein KM, Ramuzat A, Schubert B, Daum D, Neuzil P, Botman C, Castel MA, D'Onofrio A, Solomon SD, Wold N, Ruble SB. Chronic vagal stimulation for the treatment of low ejection fraction heart failure: results of the NEural Cardiac TherApy foR Heart Failure (NECTAR-HF) randomized controlled trial. Eur Heart J. 2015 Feb 14;36(7):425-33. doi: 10.1093/eurheartj/ehu345. Epub 2014 Aug 31. PMID 25176942
- [Result] De Ferrari GM, Stolen C, Tuinenburg AE, Wright DJ, Brugada J, Butter C, Klein H, Neuzil P, Botman C, Castel MA, D'Onofrio A, de Borst GJ, Solomon S, Stein KM, Schubert B, Stalsberg K, Wold N, Ruble S, Zannad F. Long-term vagal stimulation for heart failure: Eighteen month results from the NEural Cardiac TherApy foR Heart Failure (NECTAR-HF) trial. Int J Cardiol. 2017 Oct 1;244:229-234. doi: 10.1016/j.ijcard.2017.06.036. Epub 2017 Jun 10. PMID 28663046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Start: 21-Sep-2011. First implant: 28-Sep-2011.Last Implant: 20-June-2013.
  118 patients enrolled, 96 were found to be eligible and were implanted across 24 centres (7 sites with 5-10 implants, 1 site with 13 implants).
  95 patients were randomized.
Pre-assignment Details: 22 patients were excluded after enrollment. 18 patients did not meet the inclusion criteria. 4 patients decided to withdraw their consent.
  96 patients were finally implanted with the investigational device. One patient died after implant and before randomization. Randomization was done only after the investigational device implant had occurred.
Groups:
- Therapy: Vagus nerve stimulation system was implanted in the Therapy group as well as in the control group.
  Patients were randomized in a 2 : 1 ratio to receive therapy (VNS ON, Therapy) or control (VNS OFF, Control) for a 6-month period.
  The experimental arm was receiving vagus nerve stimulation soon after implant. Patients randomized to control arm were not receiving right vagal nerve stimulation for the first 6-months post-implant, after which they did also receive therapy.
- Control: Control group was implanted with study system like the experimental arm, but did receive no therapy until 6-month cross-over.
  Vagal Nerve Stimulation System was implanted but inactive for the first 6 months after implant:
  Patients randomized to control arm did not receive right vagal nerve stimulation for the first 6-months post-implant, after which they will also receive therapy.
Period: Randomization Phase
Arm/Group | Therapy | Control
Started | 63 (The randomization phase of the study started after implant of the investigational device system.) | 32 (The randomization phase of the study started after implant of the investigational device system.)
Completed | 62 (The study randomization phase ended after all patients have had their 6 month follow-up visit.) | 30 (The study randomization phase ended after all patients have had their 6 month follow-up visit.)
Not Completed | 1 | 2
Not completed — Death | 1 | 2
Period: 6-18 Month All VNS Active
Arm/Group | Therapy | Control
Started | 62 (Primary Study Phase ended with completion of the 18 months follow-up visit for the last patient) | 30 (Primary Study Phase ended with completion of the 18 months follow-up visit for the last patient)
Completed | 58 | 27
Not Completed | 4 | 3
Not completed — Death | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Heart Transplant | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients had a documented LVejection fraction (LVEF) of ≤ 35%, an LV end diastolic dimension (LVEDD) of ≥55 mm, and a New York Heart Association (NYHA) classification of II or III. Patients also had been treated with medical therapy per European heart failure guidelines for at least 30 days prior to enrolment.
Groups:
- Therapy: Therapy group was implanted with study system like the control arm, but did receive therapy soon after implant
- Control: Control group was implanted with study system like the experimental arm, but will receive no therapy until 6-month cross-over.
  Vagal Nerve Stimulation System was implanted but inactive for the first 6 months: Patients randomized to therapy arm with receive right vagal nerve stimulation. Patients randomized to control arm will not receive right vagal nerve stimulation for the first 6-months post-implant, after which they will also receive therapy.
- Total: Total of all reporting groups
Arm/Group | Therapy | Control | Total
Number analyzed (Participants) | 63 | 32 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (12.2) | 59.3 (10.1) | 59.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 56 | 26 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 13 | 6 | 19
  Czech Republic | 6 | 4 | 10
  Belgium | 1 | 1 | 2
  United Kingdom | 12 | 4 | 16
  Italy | 5 | 5 | 10
  France | 4 | 3 | 7
  Germany | 12 | 4 | 16
  Spain | 10 | 5 | 15
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (5.9) | 31.2 (5.1) | 29.9 (5.5)
Loop diuretics [Count of Participants; unit: Participants] | 54 | 32 | 86
Statin [Count of Participants; unit: Participants] | 50 | 19 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End-systolic Dimension (LVESD)
Description: Change in the Left ventricular end-systolic dimension (LVESD) between Baseline and the value at the end of the randomization phase (6 months after Baseline) i.e. 6 months after vagus nerve stimulation in the THERAPY Arm. No Vagus nerve stimulation during that time window in the CONTROL Arm.
  The sign (- ) indicates a reduction in the LVESD. Minus means a reduction in LVESD.
  The change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline).
Time Frame: LVESD at Baseline and at 6-months post Baseline
Population: The sign (- ) indicates a reduction in the LVESD. Participants without paired endpoint data did not contribute to the analysis.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Therapy: Vagus nerve stimulation system was implanted. Patients were randomized in a 2 : 1 ratio to receive therapy (VNS ON) or control (VNS OFF) for a 6-month period.
  The experimental arm was receiving vagus nerve stimulation starting at Baseline.
- Control: Control group was implanted with study system like the experimental arm, but did not receive vagus nerve stimulation for the first 6 months after Baseline, after which they will also receive vagus nerve stimulation.
  Vagal Nerve Stimulation System was implanted but inactive for the first 6 months.
Arm/Group | Therapy | Control
Number analyzed (Participants) | 59 | 28
cm | -0.04 (0.25) | -0.08 (0.32)

2. Primary Outcome: Percentage of Surviving Participants
Description: As pre-specified in the study protocol, the All-cause Survival endpoint combined both groups into one analysis population. Subjects contributed data according to the follow-up period during they received VNS therapy (Implant through 18 months for Therapy subjects, 6 through 18 months for Control subjects). Control patients who exited the study in the first 6 months, or who did not have a 6 month visit, were excluded.
Time Frame: 18-months
Population: Therapy group received VNS from implant to 18 months. Control group received VNS from 6 months to 18 months. These follow-up periods contributed to the endpoint analysis. Both groups were combined for mortality endpoint analysis. Control patients who exited the study in the first 6 months, or who did not have a 6 month visit, were excluded.
Measure: Number (90% Confidence Interval); unit: Percentage of participants surving
Groups:
- All Patients in Active VNS Periods: All patients in VNS active study periods. Therapy 0-18 months and Control 6-18 months.
Arm/Group | All Patients in Active VNS Periods
Number analyzed (Participants) | 92
Percentage of participants surving | 95 [91 to 99]

3. Secondary Outcome: LVEF, Left Ventricular Ejection Fraction
Description: LVEF, left ventricular ejection fraction.
Time Frame: LVEF at Baseline and at 6-months after Baseline
Population: LVEF echocardiographic measurements were made at Baseline and at 6 months after Baseline. Participants without paired endpoint data did not contribute to the analysis.
Measure: Mean (Standard Deviation); unit: % of blood ejected from ventricle
Groups:
- Control: Control group was implanted with study system like the experimental arm, but did not receive vagus nerve stimulation for the first 6 months after Baseline, after which they also did receive vagus nerve stimulation.
  Vagal Nerve Stimulation System was implanted but inactive for the first 6 months.
Arm/Group | Therapy | Control
Number analyzed (Participants) | 59 | 27
% of blood ejected from ventricle
  Baseline | 30.5 (6.0) | 30.8 (4.2)
  6 months after Baseline | 32.7 (6.4) | 32.1 (5.6)

4. Secondary Outcome: Exercise Capacity, Peak VO2
Description: Assessment of functional capacity (e.g., peak VO2) as measures related to patient heart failure status.
Time Frame: Measurements at Baseline and at 6-months after Baseline
Population: Participants without paired endpoint data did not contribute to the analysis.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Control: Control group was implanted with study system like the experimental arm, but did not receive vagus nerve stimulation for the first 6 months after Baseline, after which they did also receive vagus nerve stimulation.
  Vagal Nerve Stimulation System was implanted but inactive for the first 6 months.
Arm/Group | Therapy | Control
Number analyzed (Participants) | 56 | 27
ml/kg/min
  Baseline | 15.6 (3.9) | 15.2 (3.3)
  6 months after Baseline | 15.8 (4.4) | 14.7 (3.6)

5. Secondary Outcome: LVESV, Left Ventricular End Systolic Volume
Description: Measurements of LVESV, left ventricular end systolic volume at Baseline and 6 months after Baseline in the Control Arm and in the Therapy Arm
Time Frame: At Baseline and at 6-months after Baseline
Population: Measurements of LVESV, left ventricular end systolic volume at Baseline and at 6-months after Baseline. Participants without paired endpoint data did not contribute to the analysis.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Control: Control group was implanted with study system like the experimental arm, but did not receive vagus nerve stimulation for the first 6 months after Baseline, after which they did also receive vagus nerve stimulation.
  Vagal Nerve Stimulation. System was implanted but inactive for the first 6 months.
Arm/Group | Therapy | Control
Number analyzed (Participants) | 59 | 27
ml
  Baseline | 154.7 (58.5) | 164.0 (39.2)
  6 months after Baseline | 142.5 (57.1) | 152.1 (43.8)

ADVERSE EVENTS:
Time Frame: Adverse events information collected during the randomization phase, (6 month) is referred to. During this time period the primary efficicacy endpoint measurements were done and information collected. Only during these initial 6 months there were two goups of patients. After 6 month all patients had received vagus nerve stimulation. An additional Arm/Group ("All Patients - 6 to 18 Months" ) was added to present AEs collected from end of randomization phase until end of safety endpoint period.
Description: Adverse Event Definitions as per ISO 14155 were utilized. The study had only patients from European countries enrolled.
Groups:
- Therapy: Vagus nerve stimulation system was implanted in the Therapy group as well as in the control group.
  Patients were randomized in a 2 : 1 ratio to receive therapy (VNS ON, Therapy) or control (VNS OFF, Control) for a 6-month period.
  Patients randomized to therapy arm were receiving right vagal nerve stimulation shortly after implant.
- Control: Control group was implanted with study system like the experimental arm, but did receive no therapy until 6-month cross-over.
  Patients randomized to control arm did not receive right vagal nerve stimulation for the first 6-months post-implant, after which they did also receive therapy.
- All Patients - 6 to 18 Months: All patients were receiving vagus nerve stimulation after the initial 6 months of randomization.
  Three of the initially 95 randomized patients died before the end of the randomization phase, reducing the number to 92 patients.
  Note, 5 patients did not complete the Randomization phase with the 6 month follow up visit, but were still participating in the study at the time the Randomization Phase Analysis was done. These 5 patients were at risk to have an AE and were included in this analysis set (N=92)
Arm/Group | Therapy | Control | All Patients - 6 to 18 Months
All-Cause Mortality (participants affected / at risk) | 1/63 | 2/32 | 3/92
Serious Adverse Events (participants affected / at risk) | 21/63 | 18/32 | 44/92
Other Adverse Events (participants affected / at risk) | 32/63 | 15/32 | 66/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapy (N=63) | Control (N=32) | All Patients - 6 to 18 Months (N=92)
HF hospitalization, anticipated (Cardiac disorders) | 7 (10) | 5 (9) | 18 (32) — anticipated Heart Failure hospitalizations
Cardiovascular - Non Heart Failure, anticipated (Cardiac disorders) | 7 (9) | 5 (7) | 16 (26) — anticipated Cardiovascular Serious Adverse events, which were not related to Heart Failure
Pulmonary Serious Adverse Events, anticipated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 5 (6) — anticipated Pulmonary Serious Adverse Events
Genitourinary, anticipated (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (2) — anticipated Genitourinary Serious Adverse Events
Other Non Cardiocascular, anticipated (General disorders) | 7 (7) | 7 (7) | 22 (33) — Other anticipated Non Cardiocascular serious adverse events
Investigational device system related, anticipated (Product Issues) | 9 (9) | 4 (4) | 2 (2) — anticipated Investigational device system related serious adverse device effects
Heart Failure Hospitalizations, unanticipated (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) — unanticipated Heart Failure Hospitalizations
Cardiovascular - Non Heart Failure, unanticipated (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) — unanticipated Cardiovascular - Non Heart Failure
Pulmonary Serious Adverse Events, unanticipated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) — unanticipated Pulmonary Serious Adverse Events
Genitourinary, unanticipated (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) — unanticipated Genitourinary
Investigational device system related, unanticipated (Product Issues) | 0 (0) | 0 (0) | 1 (1) — unanticipated Investigational device system related
Other Non Cardiocascular, unanticipated (General disorders) | 0 (0) | 0 (0) | 0 (0) — Other unanticipated Non Cardiocascular
Death, anticipated (Cardiac disorders) | 1 (1) | 2 (2) | 3 (3) — anticpated death due to any cause
Death, unanticipated (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) — Death, unanticipated, due to any cause
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapy (N=63) | Control (N=32) | All Patients - 6 to 18 Months (N=92)
Cardiovascular HF related, anticipated (Cardiac disorders) | 15 (20) | 7 (9) | 21 (31) — anticipated Cardiovascular Heart Failure related non serious adverse events
Cardiovascular - not HF related, anticipated (Cardiac disorders) | 21 (31) | 13 (18) | 28 (40) — anticipated Cardiovascular - not Heart Failure related adverse events
Pulmonary non serious adverse events, anticipated (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 8 (8) — anticipated Pulmonary non serious adverse events (non-cardiovascular)
Genitourinary, anticipated (Renal and urinary disorders) | 1 (1) | 1 (2) | 3 (3) — Genitourinary non - serious, anticipated
Other Non-cardiovascular, anticipated (General disorders) | 19 (28) | 13 (20) | 34 (56) — Other Non-cardiovascular non-serious adverse events, anticipated
Investigational System-Related anticipated (Investigations) | 32 (55) | 11 (18) | 25 (34) — Investigational System-Related non-serious adverse events, anticipated
Cardiovascular HF related, unanticipated (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) — unanticipated Cardiovascular HF related non-serious adverse events
Cardiovascular - not HF related, unanticipated (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) — Cardiovascular - not HF related, unanticipated
Pulmonary non serious adverse events, unanticipated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) — Pulmonary non serious adverse events, unanticipated
Genitourinary, unanticipated (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) — Genitourinary, unanticipated non serious
Other Non-cardiovascular, unanticipated (General disorders) | 0 (0) | 0 (0) | 0 (0) — Other Non-cardiovascular, unanticipated
Investigational System-Related unanticipated (Product Issues) | 0 (0) | 0 (0) | 0 (0) — Investigational System-Related unanticipated

LIMITATIONS AND CAVEATS:
Inappropriate patient selection may have also contributed to the neutral findings. In the present study, therapy patients experienced side effects (e.g. neck pain, coughing), which limited programming to low stimulation amplitudes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No